CLINICAL TRIAL: NCT00799292
Title: Effects of Cervical Vasopressin Versus no Premedication on Blood Loss During Vaginal Hysterectomy
Brief Title: Comparison of the Effects of Cervical Vasopressin Versus no Premedication on Blood Loss During Vaginal Hysterectomy: A Randomized, Placebo Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ascher-Walsh, Charles, M.D. (Individual)
Responsible Party: Charles Ascher-Walsh MD, MPH, Mt Sinai School of Medicine, Department of Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASW 123
Record Dates: First submitted 2008-10-21; First posted 2008-11-27 (Estimated); Results first posted 2008-11-27 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2008-11

CONDITIONS: Blood Loss During Vaginal Hysterectomy
MeSH Terms: interventions — Vasopressins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No injection (No Intervention): Patients did not receive an injection at cervix prior to beginning the procedure
- Injection of vasopressin (Experimental): Patients will be randomized to receive 20cc of dilute vasopressin (20units in 50cc normal saline)injected at cervix at beginning of the hysterectomy
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — 20cc of dilute vasopressin (20units in 50cc normal saline). At beginning of the procedure 5cc injected were injected at 2,4,8 and 10 o'clock on the cervix
  Arms: Injection of vasopressin

SUMMARY:
Vasoconstrictive agents are increasingly being used in order to decrease blood loss during vaginal hysterectomy. The first reported study of the use of a vasoconstrictive agent for this purpose was on the use of epinephrine injected intracervically preoperatively by England, et. al. They demonstrated a significant decrease in the amount of blood lost during the surgery but also demonstrated a significant increase in the risk of post-operative infections, most frequently a vaginal cuff cellulitis requiring antibiotic treatment. Recent studies using vasopressin as the vasoconstrictive agent have also found the same significant decrease in blood loss while not demonstrating a difference in the rate of post-operative infections. The more recent studies by Speer and Unger , and Kammerer-Doak, et.al. were larger, better designed studies and are considered more credible. More surgeons are therefore injecting vasopressin intracervically preoperatively.

Some surgeons believe that the injection of vasopressin intracervically prior to the initial incision of a vaginal hysterectomy effects surgical plains and therefore makes the surgical dissection more difficult. This is thought to possibly both add to operative time and increase the rate of complications. The aforementioned studies used the injection of saline as a control for the injection of vasopressin or epinephrine. To date, no study has compared the use of vasopressin versus no injection in a controlled, randomized manner. We do not know if the injection of saline intracervically may actually increase the amount of bleeding over the baseline and therefore the decreased blood loss caused by the injection of vasopressin my actually be overestimated.

We propose to compare the effects of injecting vasopressin intracervically preoperatively versus no preoperative medication. We will not only evaluate the amount of operative blood loss, but also compare operative time and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* women greater that 18 undergoing vaginal hysterectomy for any indication, with or without concomitant procedures

Exclusion Criteria:

* women with a significant medical condition, including severe liver disease, congestive heart failure, documented coronary artery disease, impaired renal function determined by an elevated serum creatinine, asthma with steroid use in the past year, and migraines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, MPH, Principal Investigator — Mt Sinai School of Medicine, Dept Obstetrics and Gynecology
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Ascher-Walsh CJ, Capes T, Smith J, Michels A. Cervical vasopressin compared with no premedication and blood loss during vaginal hysterectomy: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):313-8. doi: 10.1097/AOG.0b013e3181954c44. PMID 19155900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment and informed consent was obtained prior to the operation in the gynecology clinic or private offices from 1/2004 - 1/2005.
Pre-assignment Details: Randomization occurred at the time of surgery.
Groups:
- Injection of Vasopressin: Patients will be randomized to receive 20cc of dilute vasopressin (20 units in 50cc normal saline) injected at cervix at beginning of the hysterectomy.
Period: Overall Study
Arm/Group | No Injection | Injection of Vasopressin
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Injection | Injection of Vasopressin | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Blood Loss During Vaginal Hysterectomy
Time Frame: Blood loss will be assessed at the end of the operative procedure
Reporting Status: Not Posted

2. Secondary Outcome: Operative Time and Complication Rates
Time Frame: Duration of procedures and immediate post-operative stay in hospital
Reporting Status: Not Posted

3. Primary Outcome: Estimated Blood Loss
Description: Estimated blood loss as mL
Time Frame: Duration of vaginal hysterectomy
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | No Injection | Injection of Vasopressin
Number analyzed (Participants) | 29 | 29
mL | 266.4 (240.50) | 145.3 (137.14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No